CLINICAL TRIAL: NCT07352462
Title: Volatile Organic Compounds Analysis for Rapid Testing Using EXhaled Breath for Respiratory Infection in Hospitalised Patients
Brief Title: Volatile Organic Compounds Analysis by GC-MS for Diagnostic of Hospitalised Patients With Respiratory Infections Using Exhaled Breath
Acronym: VORTEX-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL25_0600; 2025-A01544-45 (Other: ID-RCB)
Record Dates: First submitted 2025-11-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Infections; COVID-19; Influenza Virus Infection; Legionella Pneumophila Infections
Keywords: Pandemic preparedness; Volatilome; Breath research; Respiratory infections; Diagnosis
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19; Legionnaires' Disease; Disease

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional diagnostic study using case-control sampling, where the number of cases and non-cases is fixed in advance, and a gold standard comparison is used. 0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bacterial respiratory infection (Experimental): To classify patients, an adjudication committee will base its decision on a range of clinical and biological factors:
  * The ICD-10 code (International Classification of Diseases, 10th revision) assigned to the patient during their treatment
  * Radiological examination indicating bacterial pneumonia (community-acquired pneumonia or CAP)
  * Biological results:
    * Microbiological diagnostic tools (RT-PCR tests, culture) indicating a bacterial infection.
    * Procalcitonin measurement (indicating a bacterial infection if > 0.1 µg/L)
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using GC-MS
- Viral respiratory infection (Experimental): To classify patients, an adjudication committee will base its decision on a range of clinical and biological factors:
  * The ICD-10 code (International Classification of Diseases, 10th revision) assigned to the patient during their treatment
  * Radiological examination not indicating bacterial pneumonia
  * Biological results:
    * Microbiological diagnostic tools (RT-PCR tests, culture) indicating a viral infection. For example, respiratory infections will be attributed to a virus if at least one of the diagnostic tests used is positive for a virus or if the interferon test shows a very high score.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using GC-MS
- Undetermined respiratory infection (Experimental): All patients who matched the inclusion criteria and could not be classified into groups 1 or 2 by an adjudication committee.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using GC-MS
- Healthy patients (Placebo Comparator): The group of healthy volunteers, serving as the control group, will be composed of adult subjects with no respiratory symptoms or known acute or chronic pathology at the time of inclusion. They will be sampled using the same methods as the other groups in order to enable a reliable comparison of the metabolic signatures obtained.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using GC-MS

INTERVENTIONS:
Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using GC-MS — The collection and analysis of exhaled air for VOC detection is a non-invasive, painless procedure carried out offline. It can be summarised as follows:
  1. Collection of 0.5-1 litre of exhaled air in a single-use Tedlar® bag
  2. Transfer the exhaled air sample to a thermodesorption tube. The thermodesorption tube will be sent to the laboratory responsible for the analysis within 1-5 days of collection.
  3. The breath sample will be analysed in the laboratory using thermal desorption-GC/MS.
  4. Processing of the raw data to determine the chemical composition of VOCs and identify the compounds present in the exhaled air sample.
  5. Statistical analysis of all generated data will be performed to identify interesting VOC profiles.

SUMMARY:
Emerging respiratory diseases represent a global threat. Viruses such as influenza and coronaviruses have been the main drivers of pandemics over the past century. More broadly, the impact of these respiratory infections is not limited to pandemic risks. Indeed, some of them also trigger seasonal epidemics with a significant medical and economic burden. Consequently, it is essential to strengthen global surveillance, and diagnostic capacities for the pathogens responsible for respiratory infections.

The diagnosis of respiratory infections is even more important in cases of severe infection, as it helps guide and adapt patient management according to the responsible pathogen.

A promising and well-recognized approach is the analysis of exhaled breath, which contains a complex mixture of volatile organic compounds (VOCs), also known as the "volatilome." The volatilome is influenced by the patient's metabolism, immune system, and microbiome, and can be disrupted by the presence of a pathogen.

A parallel clinical study, VORTEX-1, aims to establish the performance of breath analysis for the diagnosis of respiratory infections in the context of the general population, or patient triage in emergency wards. This study targets patients with non-severe respiratory infections, mostly caused by viral pathogens.

Thanks to a specific technique, the VORTEX-1 study will make it possible to test a direct on-site sampling and analysis process, painless and with real-time chemical detection.

This methodology, highly suited to triage situations, remains difficult to apply in the case of respiratory infections requiring hospitalization. Indeed, hospitalized patients are usually admitted to different units depending on their clinical status, risk factors, or bed availability. This diversity of settings makes it impossible to implement a process that depends on an instrument which cannot be available or moved in real time across all units. To address this challenge, the investigators will use an alternative method.

In the VORTEX-2 trial, samples of exhaled gases will be collected directly at the patient's bedside using a single-use device for breath collection. The samples will then be transferred to a laboratory for analysis. This approach is more suitable for severe respiratory infections.

To be as comprehensive as possible in the study of the volatilome in the context of respiratory infections, it is important to include hospitalized patients and to develop a system that can also be implemented in routine clinical practice.

The link between the two studies (VORTEX-1 and VORTEX-2) will be established through a "control" group, consisting of healthy subjects (without respiratory infections or severe/chronic diseases), whose breath will be collected using both approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Having signed a written informed consent
* Presenting a NEWS-2 score of 5 (>4) or one of the individual score criteria rated 3
* Hospitalized in one of the HCL (Hospices Civils de Lyon) departments participating in the study
* With clinical signs of acute respiratory infection, or with a clinical presentation of acute community-acquired pneumonia, nasopharyngitis, angina or laryngitis (except for healthy patients)

Exclusion Criteria:

* Healthy volunteers:
* Age: < 18 years
* Alcohol consumption less than 12 hours
* Person with co-morbidities such as chronic respiratory failure, type II diabetes, cancerous processes, chronic liver disease, chronic kidney disease
* Clinical signs of acute respiratory infection
* Persons who are unable to blow into exhaled-air analysis devices (in accordance with instructions for use)
* Persons under legal protection
* Pregnant women, women in labor or nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Patients with respiratory symptoms
* Age: < 18 years
* Patients whose symptoms have been present for more than 7 days
* Persons unable to blow into the device for breath analysis (in accordance with the operating instructions)
* Patients suffering from cystic fibrosis
* Patients with severe chronic respiratory insufficiency requiring long-term oxygen therapy or NIV (non-invasive ventilation), excluding CPAP (Continuous Positive Airway Pressure) for sleep apnea
* Patients under legal protection
* Pregnant women, women in labor or nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 777 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-02-03 (Estimated)

PRIMARY OUTCOMES:
Description of the breath composition based on the area under each peak of exhaled air according to three levels of classification | day one
  Levels of classification :
  * Patients with bacterial or viral respiratory infection vs. no respiratory infection (healthy subjects = control group)
  * Patients with viral vs. bacterial respiratory infection vs. undetermined respiratory infection vs. healthy subjects
  * Patients with respiratory infection due to Legionella spp vs another bacterium vs SARS-CoV-2 vs influenza vs another virus vs undetermined respiratory infection vs healthy subjects

SECONDARY OUTCOMES:
Comparison of the overall properties of the test on exhaled air with the clinical classification of a severe respiratory infection used in practice. The test will therefore aim to differentiate patients with a respiratory infection who are hospitalized w | Day one
  Overall properties of the exhaled air test in comparison with the clinical classification of severe respiratory infection as used in practice.The test will aim to differentiate between hospitalised patients with a respiratory infection and a NEWS-2 score of over 4, and a control group of healthy patients. The overall performance of the test will be evaluated on several models, based on the area under the ROC curve (AUC) calculated from model predictions. Predicted AUCs will be compared to an expected AUC of 0.7 by bootstrapping
Differentiation of the three groups of participants-those with a viral respiratory infection, those with a bacterial respiratory infection, and healthy subjects-will be evaluated using the area under the curve (AUC), in order to assess the performance | Day one
  Evaluate the performance (same as secondary outcome 1) of the chemical analysis of exhaled air in differentiating between three groups of participants: those with a respiratory infection caused by a virus, those with a respiratory infection caused by bacteria, and healthy subjects.
Evaluation of viral load in respiratory samples will be performed by retesting all nasopharyngeal samples positive for an influenza virus, SARS-CoV-2, or Legionella. This criterion will correspond to the breath composition associated with viral load. | Day one
  The study will be based on the overall properties of the breath test compared with the clinical classification of severe respiratory infection used in practice. The test will therefore aim to differentiate between six groups. These performances will be evaluated using the AUC. The AUCs calculated from the predictions of each model developed will be compared to an expected AUC of 0.7 by bootstrap.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients'' exhaled air according to viral (influenza and SARS-CoV-2) or bacterial (Legionella) load, in order to identify biomarkers whose excretion correlates with viral and bacterial load.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients' exhaled air based on the presence of co-infection, in order to define biomarkers whose excretion is associated with these co-infections.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients' exhaled air based on innate and adaptive immune responses in patients with and without respiratory infections. Understand any classification errors due to immune responses.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the chemical analysis of exhaled air between patients with and without an impaired type I interferon response.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients' exhaled air based on the composition of the active respiratory microbiota (nasopharyngeal or pulmonary) in patients with and without respiratory infections. Understand any classification errors due to the composition of the active respiratory microbiota.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients' exhaled air based on the value of the NEW2 score at inclusion.
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of patients' exhaled air based on three clinical progression groups: worsening, stagnation or improvement based on changes in the clinical score (NEW2).
Description of the breath composition based on the AUC of each peak | Day one
  Analyse and describe the composition of healthy volunters' exhaled air based on online analysis process (VORTEX-1 clinical study) and the offline analysis process (VORTEX-2 clinical study).

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Emergency department (Hôpital de la Croix-Rousse, Hospices Civils de Lyon), Lyon
  - Infectious Disease Service of Hôpital de la Croix-Rousse (Hospices Civils de Lyon), Lyon
  - Intensive Care Unit of Hôpital de la Croix-Rousse (Hospices Civils de Lyon), Lyon
  - Intensive Care Unit of Hôpital Lyon Sud (Hospices Civils de Lyon), Lyon
  - Internal Medecine Unit of Hôpital de la Croix-Rousse (Hospices Civils de Lyon), Lyon
  - National reference center for respiratory viruses (Hôpital de la Croix-Rousse, Hospices Civils de Lyon), Lyon
  - Pneumology Unit of Hôpital de la Croix-Rousse (Hospices Civils de Lyon), Lyon

IPD SHARING:
Plan to Share IPD: No